CLINICAL TRIAL: NCT02072616
Title: Detection of Circulating Tumor Cells for the Diagnostic of Pancreatic Adenocarcinoma.
Acronym: CTC-Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2013/0141/HP
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Circulating Tumor Cells; Pancreatic Adenocarcinoma; Circulating Tumor DNA (KRAS); CA 19.9
Keywords: Circulating Tumor Cells; pancreatic adenocarcinoma; circulating tumor DNA (KRAS); CA 19.9
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sample for Circulating Tumoral Cells (Experimental): Sampling of Circulating Tumoral Cells will be done after Pancreatic adenocarcinoma diagnosis
  Interventions: Other: Pancreatic adenocarcinoma diagnosis

INTERVENTIONS:
Other: Pancreatic adenocarcinoma diagnosis

SUMMARY:
Histological proof is a crucial and necessary step for appropriate care in oncology. In the case of pancreatic cancer, histological proof from pathological analysis of the surgical specimen is very rare due to the limited number (15-20 %) of localized tumor accessible to surgical resection. In most cases, invasive endoscopic explorations are necessary for histological diagnosis before deciding of the most appropriate treatment (palliative chemotherapy or radiochemotherapy). The endoscopic ultrasound with fine needle aspiration (EUS-FNA) is currently considered as the first-line endoscopic procedure for the cytological diagnosis of solid pancreatic tumors. The technique is performed under general anesthesia with sensitivity for the diagnosis of adenocarcinoma of 80% in case of a single procedure and 92% in situations where three different procedures are required. EUS-FNA has to be performed by a physician properly trained for this type of interventional endoscopy. Some severe complications may occur but are relatively rare in expert centers (bleeding, perforation, complications of general anesthesia ...).

Diagnostic alternative approach is biological with research in the peripheral blood of markers of tumor disease. It is possible to detect indirect markers which are molecules produced by tumor tissue (eg CA19.9) and direct markers which reflect the presence of tumor biological material (circulating tumor cells (CTCs) or circulating tumor DNA).

The value of detection of CTCs is not determined for the diagnostic and therapeutic management of pancreatic cancer. Indeed, no study has evaluated the diagnosis performance of circulating markers with EUS-FNA, the reference method for the diagnosis of unresectable forms.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, and > 18 years of age
* Patient has a nonmetastatic solid pancreatic tumor (proved by CT thoraco-abdomino-pelvic) without histological evidence
* Patient is referred for surgical treatment or biliopancreatic endoscopic ultrasound with fine needle aspiration (EUS-FNA) of a pancreatic mass
* Patient has agree to participate by giving written informed consent

Exclusion Criteria:

* metastatic pancreatic tumor
* cancer or other hematologic malignancy during treatment or in remission for less than 5 years.
* minor patient under 18 years
* contraindication to surgical treatment or contraindication to the biliopancreatic EUS-FNA
* patient under guardianship
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
sensitivity of circulating tumor cells for the diagnostic of pancreatic adenocarcinoma | Day 1
  Ratio between the numbers of patients for which CTCs were observed and patients with pancreatic adenocarcinoma confirmed by pathology (FNA OR surgical specimen)

SECONDARY OUTCOMES:
diagnostic performance of the circulating tumor DNA detection (KRAS) for the diagnosis of pancreatic adenocarcinoma | Day 1
  Sensitivity, specificity and diagnostic accuracy of the detection of circulating tumor DNA (KRAS mutation) for the diagnosis of pancreatic adenocarcinoma.
prognostic impact of circulating tumor cells and / or circulating tumor DNA (KRAS) and / or CA19.9 | Day 1
  Sensitivity, specificity and diagnostic accuracy of the combined detection of CTCs and circulating tumor DNA (KRAS mutation) for the diagnosis of pancreatic adenocarcinoma
Time to first recurrence or death | Month 36
  Time to first recurrence or death according to CTC and / or circulating tumor DNA and / or CA19.9
Time to first recurrence or death | Month 18
  Time to first recurrence or death according to CTC and / or circulating tumor DNA and / or CA19.9

CONTACTS AND LOCATIONS:
Overall Officials: David SEFRIOUI, MD, Principal Investigator — UH Rouen
Locations (1):
- UH Rouen, Rouen, France